CLINICAL TRIAL: NCT00233402
Title: A Randomized, Comparative, Controlled Phase III, Multicenter Study of Hexvix Fluorescence Cystoscopy and White Light Cystoscopy in the Detection Of Papillary Bladder Cancer and the Early Recurrence Rate in Patients With Bladder Cancer
Brief Title: Study to Improve Detection and Early Recurrence Rate in Bladder Cancer Patients Using Hexvix Fluorescence Cystoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PC B305/02; NCT00209157 (obsolete NCT alias)
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-08

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Hexvix; Fluorescence; Cystoscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard White Light Cystoscopy (Active Comparator)
  Interventions: Procedure: Standard white light cystoscopy
- Standard White Light and Hexvix Fluorescence Cystoscopy (Experimental)
  Interventions: Drug: Hexvix; Procedure: Standard white light cystoscopy

INTERVENTIONS:
Drug: Hexvix — Single Instillation, Transurethral Resection of the Bladder
  Arms: Standard White Light and Hexvix Fluorescence Cystoscopy
Procedure: Standard white light cystoscopy

SUMMARY:
The purpose of this study is to document the additional detection of papillary bladder cancer and the reduced early recurrence due to the improved detection and resection of these tumors after Hexvix cystoscopy compared to standard cystoscopy in patients with papillary bladder cancer.

DETAILED DESCRIPTION:
In superficial bladder cancer macroscopic tumors including non-invasive papillary tumors (Ta) in the bladder are relatively easy to visualize by cystoscopic examination under white light. However, dysplasia, carcinoma in situ (CIS) or small exophytic tumors are easily overlooked. These lesions are predictive of recurrence and progression of disease, and the identification of these lesions is a crucial factor for the prognosis of the patient. The present situation with 50-75% recurrence rate show the inadequacy of white light cystoscopy for detection and resection of the lesions.

A better detection of papillary bladder cancer and early detection of CIS lesions will provide the patient with a more complete TURB, a more optimal pharmacological treatment when needed, may reduce the need for follow up cystoscopies and hopefully result in a better prognosis for the patient.

The aim of the present study is to compare Hexvix cystoscopy with white light cystoscopy in the detection of histology confirmed papillary bladder cancer in patients with papillary bladder cancer and to compare early recurrence rate after Hexvix and white light transurethral resection (TURB) with white light TURB in patients with superficial bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

The patients should be indicated for a cystoscopic examination for suspected or verified papillary bladder cancer and fulfill one or more of the following criteria:

* Patients with more than one initial bladder tumor confirmed on an outpatient cystoscopy.
* Patients having recurrence within 12 months confirmed on an outpatient cystoscopy
* Patients with more than one papillary lesion at recurrence independently of the time of the recurrence confirmed on an outpatient cystoscopy

Exclusion Criteria:

* Patients with known tumors in the prostatic urethra or distal urethra
* Gross hematuria. (Note: Gross hematuria is defined as a heavy bladder bleed resulting in marked amounts of blood in the urine, which may interfere with fluorescence cystoscopy. Where the bleed is light, the patient should not be excluded if in the investigator's opinion, rinsing during cystoscopy will alleviate the possible interference with fluorescence cystoscopy).
* Patient with porphyria.
* Known allergy to hexyl aminolevulinate hydrochloride or a similar compound.
* Participation in other clinical studies with investigational drugs either concurrently or within the last 30 days.
* Pregnant or breast-feeding (all women of child-bearing potential must document a negative serum or urine pregnancy test at screening and use the contraceptive pill or intrauterine device (IUD) during the treatments and for at least one month thereafter).
* Patients who have received BCG or chemotherapy within three months prior to the initial cystoscopy/TURB, except for a single dose of chemotherapy for prevention of seeding after resection.
* Conditions associated with a risk of poor protocol compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2005-01; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H Barton Grossman, Principal Investigator — The University of Texas, MD Anderson Cancer Center, Department of Urology
Locations (25):
- United States (15):
  - Stanford Cancer Center, Department of Urology, Stanford, California
  - V.A. Medical Center, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - South Florida Clinical Research Center, Inc., Pembroke Pines, Florida
  - The Emory Clinic, Dept of Urology, Atlanta, Georgia
  - Boston University School of Medicine, Boston, Massachusetts
  - St. Joseph Mercy Hospital- Ann Arbor, Ann Arbor, Michigan
  - Urologic Clinical Research Unit, Gonda 7102, Mayo Clinic Rochester, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Medical Center, Department of Urology, New York, New York
  - URMC, Rochester, New York
  - Urological Institute at Beachwood Cleveland Clinic, Beachwood, Ohio
  - Thomas Jefferson Medical College, Department of Neurology, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Department of Urologic Surgery, Nashville, Tennessee
  - Baylor College of Medicine, Scott Department of Urology, Houston, Texas
- AKH, Klinik für Urologie der Universität Wien, Vienna, Austria
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - CHUQ Hotel-Dieu de Quebec, Québec
- Germany (5):
  - University Clinic of Giessen, Department of Urology, Giessen
  - Klinikum der Universität München-Großhardern, Urologische Klinik und Poliklinik, München
  - Urologische Klinik München-Planegg, Planegg
  - Akadem. Lehrkrankenhaus der Uni Regensburg, Klinik für Urologie, Regensburg
  - Universitätsklinik Tuebingen, Universitätsklinik für Urologie, Tübingen
- Netherlands (2):
  - Department of Urology, Academic Medical Center, University of Amsterdam, Amsterdam
  - Department of Urology, UMC St. Radboud, Nijmegen

REFERENCES:
- [Derived] Stenzl A, Burger M, Fradet Y, Mynderse LA, Soloway MS, Witjes JA, Kriegmair M, Karl A, Shen Y, Grossman HB. Hexaminolevulinate guided fluorescence cystoscopy reduces recurrence in patients with nonmuscle invasive bladder cancer. J Urol. 2010 Nov;184(5):1907-13. doi: 10.1016/j.juro.2010.06.148. Epub 2010 Sep 17. PMID 20850152

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 814 patients were included in the study at 28 medical centers in the USA, Canada and Europe between January 2005 and September 2007.
Groups:
- Comparator: Standard White Light Cystoscopy
- Hexvix Fluorescence Cystoscopy: Standard White Light and Hexvix Fluorescence Cystoscopy
Period: Overall Study
Arm/Group | Comparator | Hexvix Fluorescence Cystoscopy
Started | 384 | 395
Completed | 280 | 271
Not Completed | 104 | 124
Not completed — No pathology data | 12 | 9
Not completed — No Ta/T1 | 89 | 94
Not completed — Lost to follow up etc | 3 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comparator | Hexvix Fluorescence Cystoscopy | Total
Number analyzed (Participants) | 361 | 365 | 726
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 114 | 122 | 236
  >=65 years | 247 | 243 | 490
Age Continuous [Mean (Standard Deviation); unit: years] | 69.6 (10.63) | 68.5 (10.68) | 69 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 87 | 164
  Male | 284 | 278 | 562

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With >= 1 Ta or T1 Tumor Detected With Blue Light and Not White Light
Time Frame: Day 0
Population: Analysis was based on ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Hexvix Group: The primary endpoint was assessed from patients randomized to the Hexvix group only
Arm/Group | Hexvix Group | White Light Group
Number analyzed (Participants) | 286 | 0
percentage of participants | 16.4 [11.2 to 22.8] |

2. Primary Outcome: Comparison of the Proportions of Patients in the White Light Cystoscopy and Hexvix Groups Who Underwent TURB for a Histologically-confirmed Ta or T1 Tumor Who Had a Recurrence ( CIS, Ta, T1 or T2-T4 Tumor) Within 9 Months.
Time Frame: 9 months
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Hexvix Group | White Light Group
Number analyzed (Participants) | 271 | 280
percentage of participants | 47.2 | 56.1

3. Secondary Outcome: Proportion of False Positive Lesions of Hexvix Cystoscopy and White Light Cystoscopy.
Description: The false detection rate for Hexvix cystoscopy was calculated as the total number of false positive lesions (i.e. lesions that were suspected with blue light but had negative histology according to the Standard of Truth central panel read) divided by the total number of lesions that were suspected with blue light (i.e., false positive divided by false positive plus true positive).
  The corresponding false detection rates were also calculated for white light cystoscopy for the two groups separately.
Time Frame: Day 0
Measure: Number (95% Confidence Interval); unit: Percetange of lesion
Arm/Group | Hexvix Group | White Light Group
Number analyzed (Participants) | 361 | 365
Percetange of lesion | 12 [10.2 to 14.3] | 10 [7.9 to 11.8]

4. Secondary Outcome: Proportion of Patients With at Least One CIS Lesion Detected With Blue Light and None Seen With White Light.
Time Frame: Day 0
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hexvix Fluorescence Cystoscopy
Number analyzed (Participants) | 41
percentage of participants | 31.7 [18.1 to 48.1]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Comparator | Hexvix Fluorescence Cystoscopy
Serious Adverse Events (participants affected / at risk) | 32/381 | 39/421
Other Adverse Events (participants affected / at risk) | 193/381 | 202/421
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Comparator (N=381) | Hexvix Fluorescence Cystoscopy (N=421)
Hematuria (Renal and urinary disorders) | 4 | 5
Urinary retention (Renal and urinary disorders) | 4 | 2
Bladder perforation (Renal and urinary disorders) | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 2 | 0
Urinary bladder hemorrhage (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1
Hemorrhage urinary tract (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Artrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 3 | 2
Coronary artery disease (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 3 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Epiglottis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pheumonia (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Beningn prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Broncospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Cystoprostatectomy (Surgical and medical procedures) | 1 | 1
Nephrouruterectomy (Surgical and medical procedures) | 0 | 1
Urinary bladder excision (Surgical and medical procedures) | 1 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Death (General disorders) | 1 | 1
Gravitational edema (General disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Alcohol withdraw syndrom (Psychiatric disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Ischemia (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Cofusional state (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Comparator (N=381) | Hexvix Fluorescence Cystoscopy (N=421)
Hematuria (Renal and urinary disorders) | 64 | 63
Dysuria (Renal and urinary disorders) | 28 | 40
Bladder spasm (Renal and urinary disorders) | 18 | 20
Urinary retention (Renal and urinary disorders) | 14 | 19
Bladder pain (Renal and urinary disorders) | 13 | 17
Pollakiuria (Renal and urinary disorders) | 8 | 16
Micturition urgency (Renal and urinary disorders) | 6 | 10
Nausea (Gastrointestinal disorders) | 15 | 17
Abdominal pain (Gastrointestinal disorders) | 11 | 12
Constipation (Gastrointestinal disorders) | 11 | 10
Urinary tract infection (Infections and infestations) | 26 | 26
Procedural pain (Injury, poisoning and procedural complications) | 19 | 28
Hypertention (Vascular disorders) | 9 | 18
Hypotention (Vascular disorders) | 9 | 2
Insomnia (Psychiatric disorders) | 12 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No